CLINICAL TRIAL: NCT03718988
Title: SWAP-MEAT: Study With Appetizing Plant Food - Meat Eating Alternatives Trial
Acronym: SWAP-MEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 48285
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Microbiome; Immune Function; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Meat Products

STUDY DESIGN:
Intervention Model Description: SWAP-MEAT is a randomized, cross-over design among 30 adults randomly assigned to one of two diet sequences. Each diet sequence will consist of two phases: the Meat phase, which will consist of participants consuming their typical diet, and the Plant Alternative phase, which will consist of participants consuming plant-based meat alternatives instead of their typical meat products, for a predominantly vegetarian diet.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat Phase first (Experimental): Participants will be asked to consume traditional meat products for 8 weeks, then switch to plant-based meat alternative products for another 8 weeks.
  Interventions: Behavioral: Meat products; Behavioral: Plant Alternative products
- Plant Alternative Phase first (Experimental): Participants will be asked to consume plant-based meat alternative products for 8 weeks, then switch to traditional meat products for another 8 weeks.
  Interventions: Behavioral: Meat products; Behavioral: Plant Alternative products

INTERVENTIONS:
Behavioral: Meat products — Traditional meat products (beef burger patties, pork sausage, etc.)
Behavioral: Plant Alternative products — Plant-based alternatives (The Beyond Burger, Beyond Sausage, etc.)

SUMMARY:
This study aims to investigate the impact of replacing meat consumption with plant-based meat alternative consumption on cardiovascular health, the gut microbiome, and metabolic status.

DETAILED DESCRIPTION:
Plant-based meat alternatives that closely emulate animal protein provide a new opportunity to decrease meat consumption worldwide. Decreasing meat consumption and shifting to a plant-based diet has been linked to improvements in physical health, including decreased risk of cardiovascular disease, metabolic syndrome, and type 2 diabetes (Kahleova, Levin, & Barnard, 2017). However, the extent to which plant-based meat alternatives specifically can modulate biomarkers of physical health, particularly TMAO and IGF-1, and the gut microbiome remain relatively unexplored. It is also largely unknown to what extent consumers can feasibly and sustainably exchange meat products for plant-based meat alternatives for extended periods of time. Plant-based meat alternatives offer a promising way to support consumers' shift to a plant-based diet, and in turn, to potentially improve levels of TMAO and IGF-1 and decrease cardiovascular risk. Thus, the investigators hypothesize that consumer levels of TMAO and IGF-1 will be improved after 8 weeks of consuming plant-based meat alternative products, as compared to 8 weeks of consuming traditional meat products.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Meat consumption (beef, pork/sausage, chicken) on average ≥ once a day
* Willing to consume meat (beef, pork/sausage, chicken) ≥ 2 times a day

Exclusion Criteria:

* Weight < 110 lb
* BMI ≥ 40
* LDL-C >190 mg/dL
* Systolic blood pressure (SBP) > 160 mmHg OR Diastolic blood pressure (DBP) > 90 mmHg
* Use of any of the following drugs/supplements within the last 2 months:

  * systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral);
  * corticosteroids (intravenous, intramuscular, oral, nasal or inhaled);
  * cytokines;
  * methotrexate or immunosuppressive cytotoxic agents;
* Chronic, clinically significant, or unstable (unresolved, requiring on-going changes to medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history, Type 1 diabetes, dialysis.
* History of active cancer in the past 3 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic excessive alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day; or > 14 drinks/week.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection, multiple sclerosis and Graves' disease.
* Regular/frequent use of smoking or chewing tobacco, e-cigarettes, cigars or other nicotine-containing products.
* Regular use of prescription opiate pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Trimethylamine N-oxide (TMAO). | Baseline and 8 weeks
  Change from baseline in TMAO at 8 weeks.

SECONDARY OUTCOMES:
Insulin-like Growth Factor-1 (IGF-1) | Baseline and 8 weeks
  Change from baseline in IGF-1 at 8 weeks.
Microbiota composition | Baseline and 8 weeks
  Change from baseline in alpha diversity at 8 weeks of each phase. We will be using number of observed sequence variants ("species") determined by standard 16S rRNA amplicon sequencing (V3-V5 region followed by DADA2 to define error-corrected sequence variants) as our primary metric of alpha diversity. Higher alpha diversity is better. The units are the # of sequence variants.
Microbiota function | Baseline and 8 weeks
  Change from baseline in composite of short-chain fatty acids (SCFA) concentration (ug/g stool: acetate + propionate + butyrate) at 8 weeks of each phase.
Total Cholesterol | Baseline and 8 weeks
  Change from baseline in total cholesterol at 8 weeks of each phase.
LDL Cholesterol | Baseline and 8 weeks
  Change from baseline in LDL cholesterol at 8 weeks of each phase.
HDL Cholesterol | Baseline and 8 weeks
  Change from baseline in HDL cholesterol at 8 weeks of each phase.
Triglycerides | Baseline and 8 weeks
  Change from baseline in triglycerides at 8 weeks of each phase.
Fasting glucose | Baseline and 8 weeks
  Change from baseline in fasting glucose at 8 weeks of each phase.
Fasting insulin | Baseline and 8 weeks
  Change from baseline in fasting insulin at 8 weeks of each phase.
Weight | Baseline and 8 weeks
  Change from baseline in weight at 8 weeks of each phase.
Waist circumference | Baseline and 8 weeks
  Change from baseline in weight at 8 weeks of each phase.
Blood pressure | Baseline and 8 weeks
  Change from baseline in blood pressure at 8 weeks of each phase.

OTHER OUTCOMES:
Satisfaction with Plant Alternative products | Baseline and 8 weeks
  Average satisfaction level with meals at 8 weeks of each phase (Meat phase compared to Plant Alternative phase) using a Likert scale.
Amount of Plant Alternative product consumption. | Baseline and 8 weeks
  Average number of daily servings of traditional meat products in Meat phase compared to average number of daily servings of Plant Alternative products in Plant Alternative phase.
Gastrointestinal symptoms | Baseline and 8 weeks
  Change from baseline in gastrointestinal symptoms, as assessed by the Gastrointestinal Symptoms Study Questionnaire at 8 weeks of each phase.
Perceived stress | Baseline and 8 weeks
  Change from baseline in perceived stress, as assessed by the PSS-10 questionnaire at 8 weeks of each phase.
Perceived cognitive function | Baseline and 8 weeks
  Change from baseline in perceived cognitive function, as assessed by the PROMIS SF v2.0 - Cognitive Function Abilities 4a and PROMIS SF v2.0 - Cognitive Function 4a questionnaires at 8 weeks of each phase.
Perceived fatigue | Baseline and 8 weeks
  Change from baseline in perceived fatigue, as assessed by the PROMIS SF v1.0 - Fatigue-4a questionnaire at 8 weeks of each phase.
Perceived overall health | Baseline and 8 weeks
  Change from baseline in perceived overall health, as assessed by the PROMIS Scale v1.2-Global Health questionnaire at 8 weeks of each phase.
Perceived well-being | Baseline and 8 weeks
  Change from baseline in perceived well-being, as assessed by the WHO Well-Being Index questionnaire at 8 weeks of each phase.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D. Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Background] Crimarco A, Springfield S, Petlura C, Streaty T, Cunanan K, Lee J, Fielding-Singh P, Carter MM, Topf MA, Wastyk HC, Sonnenburg ED, Sonnenburg JL, Gardner CD. A randomized crossover trial on the effect of plant-based compared with animal-based meat on trimethylamine-N-oxide and cardiovascular disease risk factors in generally healthy adults: Study With Appetizing Plantfood-Meat Eating Alternative Trial (SWAP-MEAT). Am J Clin Nutr. 2020 Nov 11;112(5):1188-1199. doi: 10.1093/ajcn/nqaa203. PMID 32780794
- [Derived] Ward CP, Landry MJ, Cunanan KM, Raphael KL, Dant CC, Gardner CD, Pao AC. Urinary Response to Consuming Plant-Based Meat Alternatives in Persons with Normal Kidney Function: The SWAP-MEAT Pilot Trial. Clin J Am Soc Nephrol. 2024 Nov 1;19(11):1417-1425. doi: 10.2215/CJN.0000000000000532. Epub 2024 Aug 26. PMID 39514692
- See also: Study description and results summary — https://med.stanford.edu/nutrition/research/completed-studies/SWAPMEATstudy.html

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT03718988/SAP_000.pdf